CLINICAL TRIAL: NCT00110578
Title: Safety and Antiviral Efficacy of Cellular Adoptive Immunotherapy With Autologous CD8+ HIV-Specific Cytotoxic T Cells Combined With Interleukin-2 For HIV Seropositive Individuals
Brief Title: Safety and Effectiveness of Immunotherapy With Autologous HIV-Specific CD8 Cells in HIV Infected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5U01AI054334-02 (NIH); AI54334
Record Dates: First submitted 2005-05-10; First posted 2005-05-11 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: Treatment Naive; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — aldesleukin

INTERVENTIONS:
Procedure: Adoptive transfer of HIV-specific CD8+ T cells
Drug: Aldesleukin

SUMMARY:
Effective, suppressive treatment for HIV infected patients can be a major challenge because HIV progressively destroys their immune systems. CD8 cells isolated from a patient's blood and grown in large numbers in the laboratory may increase a patient's immune system response to HIV. The purpose of this study is to determine if CD8 cells will provide effective antiviral activity against HIV when transplanted back in large numbers into HIV infected patients.

Study hypothesis: There are specific cells in the immune system that recognize and can kill HIV-infected cells.

DETAILED DESCRIPTION:
The function of CD8 cells in the human body is to kill infected target cells, such as HIV infected cells. Recent data suggest that intravenous administration of HIV-specific CD8 cells is safe, augments host immunity, and mediates a dramatic reduction in circulating HIV-infected CD4 cells. However, the observed antiviral effects are transient, and HIV infected CD4 cells re-emerge as the number of self CD8 cells declines. Augmenting CD8 cell response to HIV by immunotherapy with CD8 cells may be a useful addition to drug therapy if the infused CD8 cells can survive long-term in vivo. Administration of interleukin-2 (also known as aldesleukin or IL-2), a naturally occurring cytokine, has been proposed as a way to maintain the number of CD8 cells. This study will evaluate the safety and efficacy of immunotherapy with HIV-specific CD8 cells in HIV infected patients. Additionally, this study will determine if aldesleukin injections improve the persistence of self CD8 transplants and the duration of antiviral activity without severe toxicity.

This study will last 18 months. CD8 cells will be isolated from the blood of HIV infected patients; the cells will be allowed to multiply in the laboratory, and patients will receive back their CD8 cells. Patients will receive up to 3 infusions of self CD8 cells. On Day 0, patients will receive their first infusion of CD8 cells. On Day 7, patients will receive their second infusion of CD8 cells; this infusion will be followed by 14 days of aldesleukin administered daily by injection under the skin. Patients with less than a Grade 2 toxicity will receive a third infusion of CD8 cells; this infusion will be followed by 21 days of aldesleukin.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HIV infected
* CD4 count greater than 200 cells/mm3 at study entry
* Absolute neutrophil count greater than 1000 cells/mm3
* Willing to take Pneumocystis prophylaxis, if indicated
* Willing to comply with study requirements
* Willing to forgo other experimental therapy during the 26-week study period
* Willing to use acceptable forms of contraception

Inclusion Criteria for Treatment-Experienced Participants:

* Currently receiving treatment with an FDA-approved or expanded access antiretroviral agent (or combinations thereof) at a stable dose for at least 24 weeks prior to study entry

Inclusion Criteria for Treatment-Naive Participants:

* Have not received antiretroviral therapy for 6 months prior to study entry

Exclusion Criteria:

* Treatment with other immunomodulatory therapies (interferon, HIV vaccines, intravenous immunoglobulin), pentoxifylline, cancer chemotherapy, radiation therapy, or other investigational agents
* Past or present infection with mycobacterium avium complex, toxoplasmosis, cryptococcus, or cytomegalovirus (including retinitis)
* Active opportunistic infection at study entry or serious systemic infection requiring chronic maintenance or suppressive therapy
* Lymphoma, symptomatic visceral Kaposi's sarcoma, or any malignancy expected to require systemic therapy
* Serious psychological or emotional disorder that would affect ability to comply with study requirements or that would be exacerbated by protocol participation
* Alcohol or drug use, abuse, or dependence that, in the opinion of the investigator, would interfere with the study
* Estimated life expectancy of less than 4 months
* Abnormal neurocognitive examination
* Significant abnormality on electrocardiogram or chest radiograph
* Inability to generate CD8+ HIV-specific cytotoxic T cell clones
* Previously treated in FHCRC Protocol #827.1
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 1998-09; Study Completion 2005-04

PRIMARY OUTCOMES:
To determine the safety of administering CD8+ HIV-specific CTL clones followed by subcutaneous IL-2 (Proleukin, Chiron) daily for up to 21 days
To identify a regimen of IL-2 that will improve the in vivo persistence and function of adoptively transferred CD8+ HIV-specific CTL

SECONDARY OUTCOMES:
To determine whether the administration of IL-2 prolongs the antiviral activity of transferred CD8+ HIV-specific CTL
To determine if IL-2 promotes the accumulation of adoptively transferred CD8+ HIV-specific CTL in lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Riddell, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington (UW), Seattle, Washington

REFERENCES:
- [Derived] Chapuis AG, Casper C, Kuntz S, Zhu J, Tjernlund A, Diem K, Turtle CJ, Cigal ML, Velez R, Riddell S, Corey L, Greenberg PD. HIV-specific CD8+ T cells from HIV+ individuals receiving HAART can be expanded ex vivo to augment systemic and mucosal immunity in vivo. Blood. 2011 May 19;117(20):5391-402. doi: 10.1182/blood-2010-11-320226. Epub 2011 Mar 21. PMID 21422474